CLINICAL TRIAL: NCT02743013
Title: Clinical Pharmacology Study to Evaluate the Total Systemic Exposure and the Lung Availability of CHF 5993, Administered Via the Multi-dose Reservoir NEXThaler® Dry Powder Inhaler and Via a HFA-pressurised Metered Dose Inhaler With and Without Valved Holding Chamber, in Healthy Volunteers
Brief Title: Clinical Pharmacology Study to Evaluate the Total Systemic Exposure and the Lung Availability of CHF 5993 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-05993BA1-01; 2015-005198-19 (EudraCT Number)
Record Dates: First submitted 2016-03-31; First posted 2016-04-19 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation Spacers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- CHF 5993 100/6/12,5 pMDI (Active Comparator): with/without Charcoal Block
  Interventions: Drug: CHF 5993 100/6/12,5 pMDI
- CHF 5993 100/6/12,5 pMDI (replicate) (Active Comparator): with/without Charcoal Block
  Interventions: Drug: CHF 5993 100/6/12,5 pMDI replicate
- CHF 5993 100/6/12,5 pMDI VHC (Active Comparator): with/without Charcoal Block with Valved Holding Chamber
  Interventions: Drug: CHF 5993 100/6/12,5 pMDI with Valved Holding Chamber
- CHF 5993 100/6/12,5 DPI test 1 (Experimental): with/without Charcoal Block
  Interventions: Drug: CHF 5993 100/6/12,5 DPI Test 1
- CHF 5993 100/6/12,5 DPI test 2 (Experimental): with/without Charcoal Block
  Interventions: Drug: CHF 5993 100/6/12,5 DPI Test 2

INTERVENTIONS:
Drug: CHF 5993 100/6/12,5 pMDI
  Arms: CHF 5993 100/6/12,5 pMDI
Drug: CHF 5993 100/6/12,5 DPI Test 1
  Arms: CHF 5993 100/6/12,5 DPI test 1
Drug: CHF 5993 100/6/12,5 DPI Test 2
  Arms: CHF 5993 100/6/12,5 DPI test 2
Drug: CHF 5993 100/6/12,5 pMDI replicate
  Arms: CHF 5993 100/6/12,5 pMDI (replicate)
Drug: CHF 5993 100/6/12,5 pMDI with Valved Holding Chamber
  Arms: CHF 5993 100/6/12,5 pMDI VHC

SUMMARY:
This clinical pharmacology study is performed to evaluate the total systemic exposure and the lung availability of CHF 5993 DPI and pMDI with and without valved holding chamber, in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study related procedure.
2. Ability to understand the study procedures, the risks involved, and ability to be trained to use the pMDI device correctly with AIM™ (Aerosol Inhalation Monitor) Vitalograph®.
3. Ability to generate sufficient PIF (at least 40 L/min) using the In-Check device simulating NEXThaler® device.
4. Male and female Caucasian subjects aged 18 to 55 years inclusive.
5. Body mass index (BMI) within the range of 18 to 30 kg/m2 inclusive.
6. Non-smokers or ex-smokers who smoked < 5 pack years (pack-years = the number of cigarette packs per day, times the number of years) and stopped smoking > 1 year prior to screening.
7. Good physical and mental status, determined on the basis of the medical history and a general clinical examination, at screening and before randomization.
8. Lung function measurements within normal limits (Normal values: FEV1/FVC is > 0.70 and FEV1 > 80% predicted).
9. Female subject of non-childbearing potential (WONCBP) defined as physiologically incapable of becoming pregnant (i.e. post-menopausal or permanently sterile) and female subjects of childbearing potential (WOCBP) fulfilling one of the following criteria:

   * WOCBP with fertile male partners: they and/or their partner of childbearing potential must be willing to use a double barrier contraceptive method including one highly effective birth control method and one acceptable birth control method (male or female condom with or without spermicide and/or cap, diaphragm or sponge with spermicide), from the signature of the informed consent and until 3 months after follow-up visit;
   * WOCBP with non-fertile male partners: contraception is not required in this case.

Exclusion Criteria:

1. Blood donation (equal or more than 450 ml) or blood loss, less than 8 weeks prior screening or prior randomization.
2. Abnormal haemoglobin level defined as < 10.5 g/dl
3. For females only: pregnant and lactating female subjects, confirmed by a positive serum test at screening and/or urine test before randomization.
4. Positive HIV1 or HIV2 serology.
5. Positive results from the Hepatitis serology which indicates acute or chronic Hepatitis B or Hepatitis C.
6. Unsuitable veins for repeated venipuncture.
7. Documented history of alcohol abuse within 12 months prior to screening.
8. Documented history of drug abuse within 12 months prior to screening, or positive urine drug test performed at screening and/or before randomization.
9. Subjects who have a positive urine test for cotinine at screening and/or before randomization.
10. Clinically relevant abnormal laboratory values, suggesting an unknown disease and requiring further clinical investigation.
11. Clinically relevant and uncontrolled respiratory, cardiac, hepatic, renal, gastrointestinal, endocrine, metabolic, neurologic, or psychiatric disorder that may interfere with successful completion of this protocol.
12. Subjects with medical diagnosis of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that in the opinion of the investigator would prevent use of anticholinergic.
13. Subjects with history of asthma, including childhood asthma.
14. Known intolerance/ hypersensitivity to any of the excipients contained in any of the formulations used in the trial.
15. Abnormal 12-lead digitized Electrocardiogram (12-lead ECG) parameter (i.e.: QRS > 120 msec and/or PR > 220 msec and/or HR < 40 bpm and/or HR > 110 bpm and/or QTcF > 450 ms for males or QTcF > 470 ms for female, considering the average from triplicate) or 12-lead ECG evaluated as abnormal clinical significant by the investigator, at screening.
16. Abnormal Blood Pressure (i.e.: Diastolic Blood Pressure > 90 mmHg and/or Systolic Blood Pressure > 140 mmHg, considering the average from triplicate) at screening.
17. Participation in another clinical trial where investigation drug was received less than 8 weeks prior to screening.
18. Subject taking any drug treatment, including prescribed or OTC medicines as well as vitamins, homeopathic remedies etc, in the 14 days before the screening, with the exception of :

    1. Occasional paracetamol (maximum 2 g per day with a maximum of 10 g per 14 days for mild non-excluding conditions);
    2. Hormonal contraceptives;
    3. Hormonal replacement treatment for post-menopausal women.
19. Subject taking enzyme-inducing drugs, enzyme-inhibiting drugs, biologic drugs or any drug known to have a well-defined potential for hepatotoxicity (e.g. isoniazide, nimesulide, ketoconazole) in the 3 months before screening.
20. Heavy caffeine drinker (> 5 caffeinated beverages e.g., coffee, tea, cola per day).
21. Subject who has had a lower respiratory tract infection within 4 weeks prior to screening or prior randomization.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of the area under the curve (AUC0-t) for the systemic exposure of B17MP (active metabolite of Beclometasone Dipropionate), Formoterol and Glycopirronium Bromide. | 72 hours after adminstration
  AUC0-t
Evaluation of the Area under the curve (AUC) for the lung exposure of B17MP (active metabolite of Beclometasone Dipropionate), Formoterol and Glycopirronium Bromide after charcoal blockage. | 72 hours after adminstration
  AUC 0-t
Evaluation of the Maximum Plasma Concentration (Cmax) for the systemic exposure of B17MP (active metabolite of Beclometasone Dipropionate), Formoterol and Glycopirronium Bromide. | 72 hours after adminstration
  Cmax
Evaluation of the Maximum Plasma Concentration (Cmax) for the lung exposure of B17MP (active metabolite of Beclometasone Dipropionate), Formoterol and Glycopirronium Bromide after charcoal blockage. | 72 hours after adminstration
  Cmax

SECONDARY OUTCOMES:
Evaluate the Area Under the Curve of Beclometasone Dipropionate, B17MP (active metabolite of Beclometasone Dipropionate), formoterol and Glycopirronium bromide with and without charcoal blockage | 72 hours after adminstration
  Area Under the Curve
Evaluate the Maximum Plasma Concentration of Beclometasone Dipropionate, B17MP (active metabolite of Beclometasone Dipropionate), formoterol and Glycopirronium bromide with and without charcoal blockage | 72 hours after adminstration
  Maximum Plasma concentration
Evaluate the number of Adverse events and adverse drug reactions | 72 hours after adminstration
Evaluation of Blood pressure | 72 hours after adminstration
  Measurement of Blood pressure
Evaluation of the heart rate | 72 hours after adminstration
  Measurement of Heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- SGS CPU Antwerpen, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No